CLINICAL TRIAL: NCT05074940
Title: Phase II Study to Evaluate Amivantamab in Recurrent and Metastatic Adenoid Cystic Carcinoma
Brief Title: Amivantamab in Adenoid Cystic Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Trisha Wise-Draper (Other)
Responsible Party: Sponsor-Investigator, Trisha Wise-Draper, Principal Investigator, University of Cincinnati
Organization: University of Cincinnati (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCCC-HN-21-02
Record Dates: First submitted 2021-09-15; First posted 2021-10-12 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Salivary Gland Cancer
Keywords: Salivary Gland Cancer; Amivantamab; Adenoid cystic carcinoma
MeSH Terms: conditions — Salivary Gland Neoplasms; Carcinoma, Adenoid Cystic | interventions — amivantamab

STUDY DESIGN:
Intervention Model Description: Open-label phase II single arm trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Amivantamab (Experimental): Amivantamab weekly for the first cycle and biweekly thereafter.
  Interventions: Drug: Amivantamab

INTERVENTIONS:
Drug: Amivantamab — Patients will receive amivantamab at 1050mg weekly for the first cycle and biweekly thereafter (1400mg for patients ≥80kg).

SUMMARY:
The purpose of the study is to determine if treatment with amivantamab will be efficacious in patients with recurrent and metastatic adenoid cystic carcinoma.

DETAILED DESCRIPTION:
ACC is a rare cancer of salivary glands and other glandular tissue. It is slow growing and is usually treated with surgery and radiation. However, this type of cancer tends to have a high rate of recurrence and metastatic spread, which develops over several years. We hypothesize that amivantamab, a bispecific EGFR and MET inhibitor will be efficacious in ACC. Patients will receive amivantamab at 1050mg weekly for the first cycle and biweekly thereafter (1400mg for patients ≥80kg).

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically or cytologically confirmed adenoid cystic carcinoma. Non-salivary gland primary sites are allowed.
2. Recurrent and/or metastatic disease not amenable to other curative intent therapy. Patients must have had evidence of progressive disease by RECIST v1.1 within 6 months of study enrollment.
3. Presence of measurable disease as defined by RECIST v1.1
4. Age ≥18 years.
5. ECOG performance status, see Appendix A).
6. Patients must have adequate organ and marrow function
7. Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression in the last 4weeks.
8. Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required during the first cycle of therapy.
9. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
10. Before enrollment, a participant must be (as defined in Appendix 2: Contraceptive Guidance and Collection of Pregnancy Information)
11. A participant of childbearing potential must have a negative serum (b-human chorionic gonadotropin [b-hCG]) at screening and within 72 hours of the first dose of study treatment and must agree to further serum or urine pregnancy tests during the study.
12. A participant must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for 6 months after receiving the last dose of study drug.
13. A participant must wear a condom when engaging in any activity that allows for passage of ejaculate to another person during the study and for 6 months after receiving the last dose of study treatment. A participant who is sexually active with a partner of childbearing potential must agree to use a condom with spermicidal foam/gel/film/cream/suppository and his partner must also be practicing a highly effective method of contraception (i.e., established use of oral, injected or implanted hormonal methods of contraception; placement of an intrauterine device [IUD] or intrauterine system [IUS]). If the subject is vasectomized, they must still use a condom (with or without spermicide) for prevention of passage of exposure through ejaculation, but their partner is not required to use contraception.
14. The subject must also not donate sperm during the study and for 6 months after receiving the last dose of study drug.
15. Ability to understand and the willingness to sign a written informed consent document.
16. Participant must be willing and able to adhere to the lifestyle restrictions specified in this protocol.

Exclusion Criteria

1. History of allergy or intolerance to study drug components.
2. Prior use of amivantamab.

3 .Patients who have had chemotherapy or immunotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study. Palliative radiotherapy is allowed and does not require washout as long as it does not include a target lesion.

4. Positive hepatitis B (hepatitis B virus [HBV]) surface antigen (HBsAg) Note: Subjects with a prior history of HBV demonstrated by positive hepatitis B core antibody are eligible if they have at Screening 1) a negative HBsAg and 2) a HBV DNA (viral load) below the lower limit of quantification, per local testing. Subjects with a positive HBsAg due to recent vaccination are eligible if HBV DNA (viral load) is below the lower limit of quantification, per local testing.

5. Positive hepatitis C antibody (anti-HCV). Note: Subjects with a prior history of HCV, who have completed antiviral treatment and have subsequently documented HCV RNA below the lower limit of quantification per local testing are eligible.

6.Participant is positive for human immunodeficiency virus (HIV), with 1 or more of the following:

1. Receiving ART that may interfere with study treatment (consult sponsor for review of medication prior to enrollment)
2. CD4 count <350 at screening
3. AIDS-defining opportunistic infection within 6 months of start of screening
4. Not agreeing to start ART and be on ART>4 weeks plus having HIV viral load<400 copies/mL at end of 4-week period (to ensure ART is tolerated and HIV controlled).

7.Other clinically active infectious liver disease.

8. Participant has active cardiovascular disease including, but not limited to:

* A medical history of deep vein thrombosis or pulmonary embolism within 1 month prior to enrollment or any of the following within 6 months prior to enrollment: myocardial infarction, unstable angina, stroke, transient ischemic attack, coronary/peripheral artery bypass graft, or any acute coronary syndrome. Clinically non-significant thrombosis, such as non-obstructive catheter-associated thrombus(clots), or incidental or asymptomatic pulmonary embolism are not exclusionary.
* Participant has a significant genetic predisposition to venous thromboembolic(VTE) events such as Factor V Leiden.
* Participant has a prior history of VTE and is not on appropriate therapeutic anticoagulation as per NCCN or local guidelines.
* Uncontrolled (persistent) hypertension: systolic blood pressure >160 mm Hg;diastolic blood pressure >100 mm Hg.
* Congestive heart failure (CHF), defined as New York Heart Association (NYHA)class III-IV or hospitalization for CHF (any NYHA class; refer to Appendix 3:New York Heart Association Criteria) within 6 months of starting drug.

  9. Subject has uncontrolled illness, including but not limited to:
* Uncontrolled diabetes
* Ongoing or active infection (includes infection requiring treatment with antimicrobial therapy [participants will be required to complete antibiotics 1 week prior to starting study treatment] or diagnosed or suspected viral infection).
* Active bleeding diathesis
* Impaired oxygenation requiring continuous oxygen supplementation (e.g., due to medical condition requiring chronic continuous oxygen therapy).
* Psychiatric illness/social situation that would limit compliance with study requirements.
* Any ophthalmologic condition that is clinically unstable

  10. Active or past medical history of Interstitial lung disease (ILD)/pneumonitis, including drug-induced or radiation ILD/ pneumonitis.

  11. Participant had major surgery excluding placement of vascular access or tumor biopsy or had significant traumatic injury within 4 weeks before enrollment, or will not have fully recovered from surgery, or has surgery planned during the time the participant is expected to participate in the study. Note: Participants with planned surgical procedures to be conducted under local anesthesia may participate.

  12. Immune-mediated rash from checkpoint inhibitors that has not resolved prior to enrollment.

  13. Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1) with the exception of alopecia or Grade 2 neuropathy.

  14. Patients who are receiving any other investigational agents. Patients who have received other investigational agents previously who are no longer receiving these investigational agents may be eligible at the discretion of the PI. A 30 day washout from last dose of previous anticancer drug is required.

  15. Pregnant women are excluded from this study. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with breastfeeding should be discontinued if the mother is treated with amivantamab.

  16. Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions, and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-08-05 (Actual); Primary Completion 2025-08-05 (Estimated); Study Completion 2028-08-05 (Estimated)

PRIMARY OUTCOMES:
Overall response rate measured by RECIST criteria | 2 years
  To determine the overall response rate in patients with recurrent and metastatic adenoid cystic carcinoma treated with amivantamab.

SECONDARY OUTCOMES:
Progression free survival -measured as time of treatment allocation to confirmed progressive disease or death. | 5 years
  To determine the progression free survival and overall survival in patients with recurrent and metastatic adenoid cystic carcinoma treated with amivantamab.
Safety- measured by CTCAE v5 criteria and toxicity evaluation | 5 years
  To determine safety of amivantamab in patients with recurrent and metastatic adenoid cystic carcinoma.

OTHER OUTCOMES:
Molecular signatures of response and resistance- measured by comprehensive analysis of Transcriptome Sequencing | 2 years
  To determine the molecular signatures of response and resistance to amivantamab
Percent immune cell infiltration in responders versus non-responders, determined by IHC and/or IF | 2 years
  To determine immune cell infiltration in biopsy samples and correlation with response.
Quality of life - measured via FACT-HN | 2 years
  To evaluate the effect of amivantamab on patient quality of life using standardized patient reported outcome surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Trisha Wise-Draper, MD, PhD, Principal Investigator — University of Cincinnati
Locations (5):
- United States (5):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Rogel Cancer Center - University of Michigan Health, Ann Arbor, Michigan
  - Washington University - School of Medicine in St. Louis, St Louis, Missouri
  - University of Cincinnati Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No